CLINICAL TRIAL: NCT07168733
Title: Effect of Inspiratory Muscle Training on Diaphragm and Ab-dominal Wall Muscle Thickness With Fatty Liver Density in Elderly Women: A Randomized Controlled Trial
Acronym: IMT AND ELDERL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gümüşhane Universıty (Other)
Responsible Party: Principal Investigator, Coşkun YILMAZ, ASSOC. PROF., Gümüşhane Universıty
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2025/2; meeting date February 20, 2025 (Other: Scientific Research Ethics Committee of Istanbul Aydın University)
Record Dates: First submitted 2025-08-28; First posted 2025-09-11 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Perceived Recovery
Keywords: elderly women; health; exercise; aging; inspiratory muscle training
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Women aged 60-80 were invited to attend the laboratory on three separate occa-sions. During the initial visit, the experimental procedures were introduced and tested. Prior to the commencement of the experiment, each participant was furnished with a comprehensive explanation of the IMT procedure. Each participant underwent a week-long trial period, during which they were closely monitored by an experienced physiotherapist. The trial period involved the use of a respiratory muscle training device that was customised to meet the specific requirements of each participant. During the second visit, a series of pre-training measurements were taken and recorded. The tests included evaluations of AWMT, diaphragm thickness (DT), and (FLD), all of which were conducted under the supervision of a radiologist. After the four-week IMT training programme, final measurements were obtained during the final visit
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inspiratory muscle training (Experimental): Inspiratory muscle training group (IMT n:13) IMT was performed using the POWERbreathe® device (POWER® Breathe Classic, IMT Technologies Ltd., Birmingham, UK). The POWERbreathe® device is a pressure-threshold IMT device that provides resistance during inhalation. The user breathes in through a mouthpiece against an adjustable spring-loaded valve, which opens only when the inspiratory pressure exceeds the set threshold, thereby strengthening the inspiratory muscles over time (Kowalski & Klusiewicz, 2023). Following a one-week familiarization period, the IMT protocol was performed twice daily (morning and evening), five days per week, for four weeks. Each session consisted of 30 breathing cycles, resulting in a total of 60 cycles per day. Prior to training, the device resistance was calibrated to 40% of each participant's maximal inspiratory pressure (MIP), as reported by Çelikel et al. (2025) to promote increases in muscle size and thickness. MIP was reassessed weekly and resistance was
  Interventions: Device: Inspiratory muscle training; Other: Control
- CONTROL (No Intervention): The research group (Control Group (CG) (n:13)

INTERVENTIONS:
Device: Inspiratory muscle training — The POWERbreathe® device is a pressure-threshold IMT device that provides resistance during inhalation. The user breathes in through a mouthpiece against an adjustable spring-loaded valve, which opens only when the inspiratory pressure exceeds the set threshold, thereby strengthening the inspiratory muscles over time. Following a one-week familiarization period, the IMT protocol was performed twice daily (morning and evening), five days per week, for four weeks. Each session consisted of 30 breathing cycles, resulting in a total of 60 cycles per day. Prior to training, the device resistance was calibrated to 40% of each participant's maximal inspiratory pressure (MIP), as reported by Çelikel et al. (2025) to promote increases in muscle size and thickness. MIP was reassessed weekly and resistance was increased by 10%; progression was paused if participants experienced excessive strain.
  Arms: Inspiratory muscle training
Other: Control — The group that continues with their normal daily routines
  Arms: Inspiratory muscle training

SUMMARY:
Background: Post-menopausal estrogen decline is considered a contributing factor to sarcopenia, and inspiratory muscle training (IMT) may provide benefits in this demo-graphic. This study examined the impact of a four-week IMT program on diaphragm thickness, abdominal wall muscle thickness (AWMT; transversus abdominis, internal oblique, and external oblique), and liver fat percentage in healthy elderly women. Methods: Twenty-six women aged 60-80 years were randomly assigned to an IMT group (n = 13) or a control group (n = 13). The IMT group used the PowerBreathe® Classic device at 40% of maximal inspiratory pressure (MIP), with weekly increments of 10%. Training was performed twice daily, five days per week, with 30 breathing cycles per session (60 per day). The control group maintained their usual routines. AWMT, diaphragm thickness (DT), and fatty liver density (FLD) were measured by a radiologist before and after the intervention.

DETAILED DESCRIPTION:
1. Introduction The aging process leads to various impairments in multiple physiological systems, including the musculoskeletal and respiratory systems. One of the primary consequences of this process is the decline in overall muscle strength, which directly affects an individual's functional capacity and ability to perform daily living activities. Although this reduction in muscle mass and strength is not directly associated with any specific disease, it becomes more pronounced in elderly adults with health conditions that limit mobility. Respiratory muscle weakness alone is considered a significant limiting factor for physical fitness and may lead to clinical outcomes, including impaired lung function, reduced muscle strength, and dyspnea.

   Previous studies have reported that physical exercise provides a wide range of benefits for elderly adults, including improvements in functional capacity, reductions in infection rates, enhanced cardiovascular fitness, improved muscle fiber quality, and overall enhancements in quality of life. Aerobic exercise has been shown to exert systemic benefits, including improvements in respiratory muscle strength. Moreover, regular physical activity induces both local and systemic anti-inflammatory responses, offering protective effects against age-related chronic inflammatory pathologies (Silva et al., 2011, Can et al., 2019).

   In this context, improving respiratory function through targeted interventions is vital for maintaining independence and decreasing healthcare burdens in aging populations. In recent years, IMT has gained increasing attention due to its dual role in enhancing athletic performance and improving functional capacity in elderly adults. IMT is a resistance training approach involving moderate-intensity respiratory loading, typically at 40-60% of maximal inspiratory pressure. It is performed over short durations while yielding significant improvements in muscle strength and endurance. Home-based protocols generally consist of breathing sessions conducted twice daily, five to seven days per week.

   The practicality and safety of these home-based programs make IMT particularly suitable for elderly populations, including those with mobility restrictions. IMT has been reported to lower blood pressure in elderly adults with systolic hypertension , improve cardiac autonomic function, reduce sympathetic overactivity, and enhance vagal tone at rest in individuals with obstructive sleep apnea. Furthermore, IMT has been identified as a non-pharmacological intervention that enhances diaphragm function, supports postural balance, increases trunk stability, facilitates venous return, and ultimately reduces the risk of falls.

   With advancing age, several age-related changes occur in the respiratory system, including reduced chest wall compliance, decreased elastic recoil of the lung parenchyma, diminished respiratory muscle strength, and a blunted response to gas exchange abnormalities. These alterations are associated with decreased exercise capacity, impaired walking performance, and reduced quality of life in elderly adults. The decline in respiratory muscle function renders elderly individuals more vulnerable to disease and disability; therefore, strengthening these muscle groups is crucial for reducing the risks of morbidity and mortality. Despite this, respiratory-specific exercise strategies, such as IMT, remain underutilized in geriatric health promotion efforts.

   Although peripheral muscle exercises may yield partial gains in respiratory muscle function, more pronounced improvements have been observed when these exercises are supported with inspiratory muscle-specific training. . In the literature, the diaphragm has been reported to play an active role not only in respiratory function but also in controlling postural balance. By increasing intra-abdominal pressure, the diaphragm contributes to spinal stabilization and, in coordination with the abdominal muscles, supports balance. In this context, ultrasound imaging can be used to measure abdominal muscle thickness, and a positive correlation between muscle thickness and strength has been reported.

   Previous studies have primarily focused on the effects of IMT on respiratory per-formance, diaphragm mobility, and functional capacity in elderly populations. While these studies consistently reported improvements in inspiratory pressures and diaphragm thickness, they did not comprehensively address changes in AWMT or explore systemic outcomes such as hepatic steatosis. Furthermore, most of the available research examined either functional or structural outcomes separately, leaving a gap in understanding the dual effects of IMT on both musculoskeletal and metabolic health indicators. Our study differs from prior work in that it evaluates not only diaphragm thickness and AWMT but also liver fat density (FLD) using computed tomography in elderly women. This combined approach provides novel insight into how a short-term IMT intervention may influence both muscle structure and metabolic health. To address this gap, the present study aimed to investigate the effects of a four-week IMT intervention on diaphragm thickness and AWMT, as well as FLD, in this population. We hypothesized that IMT would lead to significant improvements in these outcomes, thereby supporting its role as a comprehensive strategy to preserve both functional capacity and metabolic health in aging women.
2. Materials and Methods 2.1. Participants This study was conducted as a parallel-group, pretest-posttest randomized con-trolled trial following the CONSORT guidelines. Before participation, all individuals received detailed information about the study and provided written informed consent following the ethical principles outlined in the Declaration of Helsinki. The study was designed following the principles of the Declaration of Helsinki and was approved by the Scientific Research Ethics Committee of Istanbul Aydın University (meeting dated February 20, 2025, number 2025/2). The sample size was calculated using G*Power software (version 3.1.9.2) based on diaphragm thickness (DT) values reported in previous studies (Holtzhausen et al., 2018), with an alpha error of 0.05, a beta error of 0.2, and a medium effect size (f = 0.25 or partial eta squared = 0.06). Considering the study design, a dropout rate of approximately 50% was anticipated. Accordingly, a sample size of 20 participants (n = 10 per group) was initially determined. However, to minimize potential issues, it was decided to include a total of 30 participants by adding 50% more participants to each group. Ultimately, four participants were excluded because they did not meet the inclusion criteria, and the study was completed with 26 participants. The two groups participating in the study consisted of healthy elderly women residing in a special care home, retired from working life, and with similar levels of sporting activity.

Inclusion criteria were defined as women aged 60-80 years (post-menopausal), who were independent in activities of daily living, demonstrated adequate cognitive function to follow instructions, had no musculoskeletal injury within the previous six months, were non-smokers, and had routine thoracic or abdominal CT images obtained for clinical indications and used in this study. Exclusion criteria included having uncontrolled cardiovascular or pulmonary disease such as heart failure or COPD/asthma exacerbation, uncontrolled hypertension, diagnosed chronic liver disease, acute respiratory infection within the last four weeks, participation in structured respiratory or resistance training within the last six months, recent thoracoabdominal surgery or hernia, use of medications known to affect muscle or liver metabolism such as systemic corticosteroids, anabolic agents, or hepatotoxic drugs, severe orthopedic or neurological conditions limiting mobility, or refusal to participate.

2.2. Experimental design Women aged 60-80 were invited to attend the laboratory on three separate occa-sions. During the initial visit, the experimental procedures were introduced and tested. Prior to the commencement of the experiment, each participant was furnished with a comprehensive explanation of the IMT procedure. Each participant underwent a week-long trial period, during which they were closely monitored by an experienced physiotherapist. The trial period involved the use of a respiratory muscle training device that was customised to meet the specific requirements of each participant. During the second visit, a series of pre-training measurements were taken and recorded. The tests included evaluations of AWMT, diaphragm thickness (DT), and (FLD), all of which were conducted under the supervision of a radiologist. After the four-week IMT training programme, final measurements were obtained during the final visit 2.3. Body composition measurement The height of participants was measured to the nearest 0.1 centimetre using a standard height meter (Seca 769, Seca, Hamburg, Germany) while standing barefoot against a wall. Body weight was measured to the nearest 0,1 kilogram using a digital scale (Beurer, model GS27). Participants' body weight was measured in kilograms (kg) without shoes and while wearing shorts and a T-shirt to minimize the influence on the results When we look at the averages of the participants in the study, for the IMT group, the age was 67.69±9.25 years, height was 159.5±4.3 cm, and weight was 70.77±3.65 kg. while for the control group, the mean age was 68±8.40 years, height was 157.85±3.05 cm, and weight was 69.46±2.22 kg.

2.4. Liver Density Analysis In this study, CT images were preferred because participants had already under-gone thoracic or abdominal CT scans as part of their routine clinical care. No additional imaging was performed for research purposes. Thus, existing clinical data were utilized, avoiding extra radiation exposure. Imaging was performed using a Siemens Somatom Definition AS 128 CT scanner during the inspiratory phase after standardized breathing instructions. Liver density was measured from a homogeneous parenchymal region without visible lesions in segment VIII adjacent to the middle hepatic vein, while diaphragm and abdominal muscle thicknesses were assessed at anatomically standardized sites. The device automatically calculated and recorded liver fat content. A liver fat value of less than 33 indicated increased hepatic steatosis.

2.5. Diaphragm Thickness (DT) Measurement Diaphragm muscle thickness measurements were obtained from computed tomography images taken for clinical reasons. The GE Revo Evo Cardiac device (Revolution EVO, Revolution Maxima, Revolution Frontier, Revolution HD, Revolution CT, GE Healthcare, WI, USA) was used for imaging. A radiologist with expertise in thoracic computed tomography performed the measurements of diaphragm muscle thickness. During the imaging procedure, the subjects were in a supine position during the deep inspiration phase. Thickness measurements were obtained at the level of the upper pole of the right kidney. The measurements were taken perpendicular to the diaphragm axis, from the midline, and the posterior line of the vertebral body. At this juncture, the diaphragm muscle was visualised and its thickness was measured.

2.6. Abdominal wall muscle thickness measurement The present study utilized data obtained from participants aged 60 and above who underwent chest or abdominal CT scans for various clinical indications. Imaging was performed using a computed tomography device, model Revo Evo of General Electric. Before undergoing imaging procedures, the participants were instructed to perform breathing exercises. On the day of imaging, participants were positioned supine on the device table. Following the completion of device settings, participants were asked to take a deep breath and hold it immediately before imaging commenced. The images under consideration were obtained during the inspiration phase. In this study, AWMT was defined as the thickness of the muscular layers of the abdominal wall (transversus abdominis, internal oblique, and external oblique), excluding subcutaneous fat and other non-contractile tissues. For simplicity, this variable is hereafter referred to as AWMT. Measurements were taken at the level of the upper iliac wings, in a plane perpendicular to the muscle plane at the level of the anterior line of the vertebral body.

2.7. Inspiratory muscle training (IMT) IMT was performed using the POWERbreathe® device (POWER® Breathe Classic, IMT Technologies Ltd., Birmingham, UK). The POWERbreathe® device is a pressure-threshold IMT device that provides resistance during inhalation. The user breathes in through a mouthpiece against an adjustable spring-loaded valve, which opens only when the inspiratory pressure exceeds the set threshold, thereby strengthening the inspiratory muscles over time. Following a one-week familiarization period, the IMT protocol was performed twice daily (morning and evening), five days per week, for four weeks. Each session consisted of 30 breathing cycles, resulting in a total of 60 cycles per day. Prior to training, the device resistance was calibrated to 40% of each participant's maximal inspiratory pressure (MIP), as reported by Çelikel et al. (2025) to promote increases in muscle size and thickness. MIP was reassessed weekly and resistance was increased by 10%; progression was paused if participants experienced excessive strain. All participants were able to complete the progressive protocol without interruption. Importantly, all IMT sessions were supervised by a licensed physiotherapist with more than five years of clinical experience in respiratory rehabilitation, who provided detailed instruction on the correct use of the POWERbreathe® device, demonstrated proper breathing techniques, and corrected participant errors during the initial sessions. Morning IMT sessions were scheduled between 8:00-10:00 a.m., while evening sessions took place between 5:00-8:00 p.m.

2.8. Statistical analysis Statistical analyses were performed using SPSS (Version 21.0 for Windows, Chicago, IL, USA), with a statistical significance level set at 0.05. The Shapiro-Wilk normality test was performed to determine the normality of the sample. The pre-test and post-test differences were determined using a Paired Samples t-test and One-Way Analysis of variance (ANOVA), with post-test and pre-test difference values used to determine between-group differences. Additionally, the effect size in the comparison of paired groups was calculated using Hedges' g It was also interpreted as follows: 0-0.19 insignificant, 0.20-0.59 small, 0.6-1.19 medium, 1.20-1.99 large, and ≥2.00 very large.

ELIGIBILITY:
Inclusion Criteria:

* were defined as women aged 60-80 years (post-menopausal), who were independent in activities of daily living,
* demonstrated adequate cognitive function to follow instructions,
* had no musculoskeletal injury within the previous six months,
* were non-smokers,
* had routine thoracic or abdominal CT images obtained for clinical indications and used in this study.

Exclusion Criteria:

* included having uncontrolled cardiovascular or pulmonary disease such as heart failure or COPD/asthma exacerbation,
* uncontrolled hypertension, diagnosed chronic liver disease,
* acute respiratory infection within the last four weeks,
* participation in structured respiratory or resistance training within the last six months,
* recent thoracoabdominal surgery or hernia, use of medications known to affect muscle or liver metabolism such as systemic corticosteroids, anabolic agents, or hepatotoxic drugs,
* severe orthopedic or neurological conditions limiting mobility, or refusal to participate.

Ages: 60 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2025-06-05 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-08-05 (Actual)

PRIMARY OUTCOMES:
pre-training | 4 week
  Assessments were performed for all participants in both groups 4 weeks before and after treatment. These parameters were assessed using pre- and post-test measurements and compared between the IMT group and the control group Diaphragm Thickness (DT)
  * Mid-diaphragm thickness (MDT)
  * Posterior diaphragm thickness (PDT)
pre-training | 4 Week
  Assessments were performed for all participants in both groups 4 weeks before and after treatment. These parameters were assessed using pre- and post-test measurements and compared between the IMT group and the control group
  -Fatty Liver Density (FLD)
pre-training | 4 week
  Assessments were performed for all participants in both groups 4 weeks before and after treatment. These parameters were assessed using pre- and post-test measurements and compared between the IMT group and the control group Abdominal Wall Muscle Thickness (AWMT)
  * Right abdominal wall muscle thickness (RAWMT)
  * Left abdominal wall muscle thickness (LAWMT)

CONTACTS AND LOCATIONS:
Locations (1):
- Gumushane Univetsity, Kelkit, Gümüşhane Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF